CLINICAL TRIAL: NCT03314480
Title: A Novel Clinical Decision Aid for the Diagnostic Management of Maxillofacial Trauma: the REDUCTION Trial - REDucing Unnecessary Computed Tomography Imaging for MaxillOfacial INjury
Brief Title: REDucing Unnecessary Computed Tomography Imaging for MaxillOfacial INjury
Acronym: REDUCTION
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Isala (Other); Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, Romke Rozema, BSc, University Medical Center Groningen
Other Study IDs: 201700304
Record Dates: First submitted 2017-10-04; First posted 2017-10-19 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Maxillofacial Injuries; Image Interpretation, Computer-Assisted; Craniocerebral Trauma; Emergency Medicine
Keywords: Multidetector Computed Tomography; Cone Beam Computed Tomography; Maxillofacial fractures; zygomaticomaxillary fractures
MeSH Terms: conditions — Maxillofacial Injuries; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midfacial fracture suspected patients: Patients who are suspected of maxillofacial fracture
  Interventions: Diagnostic Test: Standardized physical examination
- Mandibular fracture suspected patients: Patients who are suspected of a mandibular fracture
  Interventions: Diagnostic Test: Standardized physical examination

INTERVENTIONS:
Diagnostic Test: Standardized physical examination — Standarized physical examination dedicated to assess a potential fracture in the maxillofacial or mandibular region.

SUMMARY:
The aim is to prospectively assess the association between clinical parameters and the presence of maxillofacial fractures in trauma patients admitted to the emergency department. Our hypothesis is that a clinical decision aid of critical parameters reduces unnecessary produced CT scans in maxillofacial trauma patients.

DETAILED DESCRIPTION:
The REDUCTION trial is a prospective multicentre cohort study conducted at the level I emergency departments of the University Medical Center Groningen, Isala hospital (Zwolle, The Netherlands) and the level II trauma center Nij Smellinghe hospital (Drachten, The Netherlands). The increased availability of Computed Tomography (CT) in the emergency department is leading to an overuse for patients with suspected maxillofacial injury. The use of a clinical decision aid could lead to more expedient use of diagnostic imaging within this population of patients. Therefore, all maxillofacial trauma patients admitted to the emergency department are included in this trial if the consultation is within 7 days after trauma. Both maxillofacial trauma patients admitted to CT scan and patients without a radiological confirmed diagnosis are included. The research protocol was approved by the institutional review board of the University Medical Center Groningen (Groningen, The Netherlands). Informed consent was waived as patients are treated according to the standards of care. Upon admission, each patient with maxillofacial injury will be allocated as a midfacial or mandibular trauma. During physical examination, either by the emergency physician or surgical resident, a pre-defined selection of clinical parameters will be assessed focussing on the assessment of potential presence of fractures in the maxillofacial region. The standardization of this examination will be ensured using a pocket map and easy accessible online instructional video's. The clinical parameters, fracture likelihood and physical examination findings will be structurally reported in electronic health record software using a smart tool dedicated for maxillofacial injury. Data regarding patient demographics, mechanism of injury, concomitant injury, diagnostic outcome and radiation dose parameters will be derived from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* consultation within 7 days of trauma

Exclusion Criteria:

* history of maxillofacial surgery

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a maxillofacial trauma admitted to the emergency department of the cooperating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1126 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Maxillofacial fracture | Within 1 day, from admission to discharge from the emergency department
  The presence of either a maxillofacial or mandibular fracture induced by the trauma and diagnosed using CT or orthopantomography in the emergency department.

SECONDARY OUTCOMES:
Treatment outcome | Within 2 weeks upon admission to the emegency department
  The outcome of the treatment as determined by the Oral and Maxillofacial (OMF) surgeon or emergency physician classified as;
  1. Admission and direct surgical treatment
  2. Admission following elective surgery
  3. Discharge following elective surgery
  4. Discharge, expectative treatment and follow-up after seven days
  5. Discharge, conservative treatment and follow-up after seven days
  6. Discharge, conservative treatment, no follow-up

OTHER OUTCOMES:
CT time | Within 2 weeks from admission to the emergency department
  Time from admission to CT scanner
Emergency department total time of admission | Within 2 weeks from admission to the emergency department
  Total time the patient was of admitted at the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Fred KL Spijkervet, DMD PhD, Principal Investigator — University of Groningen
Locations (4):
- Netherlands (4):
  - Isala Diaconessenhuis, Meppel, Overijssel
  - Isala ziekenhuis, Zwolle, Overijssel
  - Nij Smellinghe ziekenhuis, Drachten, Provincie Friesland
  - University Medical Center Groningen, University of Groningen, Groningen

REFERENCES:
- [Derived] Rozema R, Moumni ME, de Vries GT, Spijkervet FKL, Verbeek R, Kleinbergen JYJ, Bens BWJ, Doff MHJ, van Minnen B; REDUCTION study group. A clinical decision aid for patients with suspected midfacial and mandibular fractures (the REDUCTION-I study): a prospective multicentre cohort study. Eur J Trauma Emerg Surg. 2022 Oct;48(5):4243-4254. doi: 10.1007/s00068-022-01968-1. Epub 2022 Apr 16. PMID 35430710
- [Derived] Rozema R, El Moumni M, de Vries GT, Spijkervet FKL, Verbeek R, Kleinbergen JYJ, Bens BWJ, Doff MHJ, van Minnen B; REDUCTION study group. A clinical decision aid to discern patients without and with midfacial and mandibular fractures that require treatment (the REDUCTION-II study): a prospective multicentre cohort study. Eur J Trauma Emerg Surg. 2022 Aug;48(4):2547-2558. doi: 10.1007/s00068-022-01892-4. Epub 2022 Feb 24. PMID 35211773